CLINICAL TRIAL: NCT02834260
Title: Immunosuppression During Penetrating Keratoplasty, Using a Subconjunctival Implant Releasing Dexamethasone: Tolerance and Safety Pilot Study
Brief Title: Immunosuppression During Penetrating Keratoplasty, Using a Subconjunctival Implant Releasing Dexamethasone : Tolerance and Safety Pilot Study
Acronym: IDEXACOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1608042; 2016-001168-12 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-15 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-05

CONDITIONS: Keratoconus; Fuchs' Endothelial Dystrophy; Congenital Hereditary Stromal Dystrophy of the Cornea
Keywords: absorbable implant; subconjunctival; immune rejection; safety profile; dexamethasone
MeSH Terms: conditions — Keratoconus; Fuchs' Endothelial Dystrophy; Corneal Dystrophy, Congenital Stromal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ozurdex group (Experimental): Subconjunctival injection of the absorbable implant of Dexamethasone immediately at the end of penetrating keratoplasty. The injection is made at the 12 O'Clock position is a bubble created by subconjunctival injection of balanced salt solution.
  Interventions: Drug: Dexamethasone implant OZURDEX

INTERVENTIONS:
Drug: Dexamethasone implant OZURDEX

SUMMARY:
Immune rejection episodes after penetrating keratoplasty occur in 30% of patients and constitute one of the main factors reducing graft survival. They mainly occur during the first 18 months. Prevention usually relies on a topical treatment with dexamethasone or prednisolone for standard risk patients. Eye drops are instilled three times a day during at least 3 months then tapered.

OZURDEX is an absorbable small implant that releases a total of 700 micrograms dexamethasone during several months. It is indicated for intravitreal injection to treat macular edema.

The investigators hypothesized that this implant could be used after subconjunctival injection during corneal graft, to prevent immune rejection and avoid repeated eyedrop instillations.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus
* Fuch's dystrophy
* Hereditary stromal dystrophy
* Age 18 years old and more
* Signed informed consent
* Affiliated to the French Social Security

Exclusion Criteria:

* Hypersensitivity to Dexamethasone or the excipients (polylactic and glycolic acid)
* Active ocular or periocular infection
* Advanced glaucoma
* History of herpetic or zoster keratitis
* Retinal disease for which an intravitreal injection of Ozurdex is planed for the next 3-4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
intraocular pressure | one month post graft

SECONDARY OUTCOMES:
Score of ocular discomfort | Day 1, Day 2, Day 3, Day 4, Day 5, Day 15, Month 1, Week 5, Week 6, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12
  analogic visual scale
Ocular redness | Day 1, Day 2, Day 3, Day 4, Day 5, Day 15, Month 1, Week 5, Week 6, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12
  digital picture
Rejection episodes | Day 1, Day 2, Day 3, Day 4, Day 5, Day 15, Month 1, Week 5, Week 6, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12
Graft thickness | one month post graft
Patient requiring dexamethasone eyedrops | one month post graft
Date of disappearance of the implant | up to 1 year
intraocular pressure | Day 1, Day 2, Day 3, Day 4, Day 5, Day 15, Week 5, Week 6, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12
presence of hemorrhage | Day 1, Day 2, Day 3, Day 4, Day 5, Day 15, Month 1, Week 5, Week 6, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12
  with tomography

CONTACTS AND LOCATIONS:
Overall Officials: Marie Caroline TRONE, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trone MC, Poinard S, Crouzet E, Garcin T, Mentek M, Forest F, Matray M, Thuret G, Gain P. Dropless penetrating keratoplasty using a subconjunctival dexamethasone implant: safety pilot study. Br J Ophthalmol. 2023 Feb;107(2):181-186. doi: 10.1136/bjophthalmol-2021-319376. Epub 2021 Aug 23. PMID 34426402